CLINICAL TRIAL: NCT04620395
Title: Clinical Investigation of Septic and Aseptic Prosthetic Joint Failure - Percutaneous Punch Biopsy as a Novel Way of Diagnosis Confirmation
Brief Title: Percutaneous Punch Biopsy for Diagnosis of Septic and Aseptic Prosthetic Joint Failure
Acronym: SHARP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vivantes Netzwerk für Gesundheit GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STUD.20-062; DRKS00022931 (Registry Identifier: DRKS); U1111-1257-2609 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2020-08-25; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Wear of Articular Bearing Surface of Internal Prosthetic Joint; Infection Prosthetic; Infections Joint Prosthetic; Prosthetic Joint Infection; Prosthetic Pain
Keywords: prosthetic joint; infection; wear particles; prosthetic failure; antibiotics; biopsy; joint tap
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Joint tap (No Intervention): Joint tap and aspiration of synovial fluid
- Punch biopsy (Experimental): Punch biopsy of a prosthetic joint and extraction of 5-7 biopsies from the synovial membrane
  Interventions: Diagnostic Test: Punch biopsy

INTERVENTIONS:
Diagnostic Test: Punch biopsy — A standardized biopsy kit is used for a synovial fluid tap and subsequent acquisition of up to 7 Punch biopsies through an introducer (part of the kit)
  Arms: Punch biopsy

SUMMARY:
The aim of the superiority study is to establish a reproducible, minimally invasive, cost-effective way of sample collection for microbiological and pathomorphological processing in a clinical setting with avoidance of anesthesia, multiple punctures, as well as potential deep contamination during irrigation.

DETAILED DESCRIPTION:
The main aim of the study is to demonstrate the superiority of a punch biopsy over a joint tap to rule out or prove septic prosthesis failure and thus establish a new diagnostic method. The subsequently calculated sensitivities of the previous and the procedure are used as the main indicator. In addition, we would like to prove that the total cost of diagnosing a septic / aseptic prosthesis failure using the proposed method has socio-economic advantages over the previous algorithm.

One of the secondary objectives is the evaluation of the use of a punch biopsy for simultaneous a priori pathomorphological examination of periprosthetic soft tissue samples for the determination of wear particles. Furthermore, the study is intended to demonstrate a shortening of the time span between the first suspected diagnosis of septic prosthesis failure and its reliable exclusion / detection.

ELIGIBILITY:
Inclusion Criteria:

* Preceding implantation of a shoulder, hip or knee endoprosthesis
* Acute or chronic pain in the joint
* Periprosthetic fracture
* Instability of the endoprosthesis
* Indications of wear / insufficiency of the enclosed plastic spacers
* Indications of metal abrasion
* Primary misalignment of the implant

Exclusion Criteria:

* Confirmed periprosthetic infection
* Proven allergy to fast-acting local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Improved diagnostic accuracy | up to 3 months
  Comparison of the specificity and sensibility of microbiological results for punch biopsies, the synovial fluid tap, pre-interventional blood Analysis, arthroscopic biopsies for confirmation/exclusion of a bacterial or fungal periprosthetic infection

SECONDARY OUTCOMES:
Rate of chronic periprosthetic low-grade-infections | up to 3 Months
  The incidence of hidden chronic periprosthetic infections
Correlation of microbiological results from percutaneous Punch biopsy with intraoperative findings at Revision | up to 6 Months
  Correlation of pre-revision microbiological findings and the samples taken during the endoprosthesis replacement operation, in particular the sonicate of the prosthesis and the periprosthetic membrane (gold standard for infection diagnostics)
Total Cost of Infection Diagnostics for various used methods | 1 Month
  Comparison of the respective Overall Costs for diagnostics of acute and chronic periprosthetic infections using a joint-tap, the novel punch biopsy method and arthroscopic biopsy
Rate of prosthetic failure due to wear particles | up to 1 month
  Incidence of presence of wear particles in pathomorphological examinations of the punch biopsies and the samples taken during the replacement operation
Correlation of Synovialitis score and microbiological findings | up to 2 months
  Correlation of Synovialitis score in pathomorphological examinations and microbiological verification of an acute or chronic periprosthetic infection

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Labs, PD Dr, Study Chair — Vivantes Humboldt Krankenhaus
Locations (1):
- Vivantes Humboldt-Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No